CLINICAL TRIAL: NCT00077337
Title: Phase II Trial of Depsipeptide (NSC-630176) in Colorectal Cancer Patients Who Have Received Either One or Two Prior Chemotherapy Regimens for Metastatic or Locally Advanced, Unresectable Disease
Brief Title: FR901228 in Treating Patients With Previously Treated Unresectable Locally Advanced or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000350199; SWOG-S0336
Record Dates: First submitted 2004-02-10; First posted 2004-02-12 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2005-11

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage III colon cancer; stage IV colon cancer; recurrent rectal cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — romidepsin

INTERVENTIONS:
Drug: romidepsin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as FR901228, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well FR901228 works in treating patients with unresectable locally advanced or metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the confirmed response (complete and partial) in patients with previously treated unresectable locally advanced or metastatic colorectal cancer treated with FR901228 (depsipeptide).
* Determine the time to treatment failure and overall survival of patients treated with this drug.
* Determine the qualitative and quantitative toxic effects of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive FR901228 (depsipeptide) IV over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 8 weeks until disease progression and then every 3 months until 1 year after study entry and then every 6 months until 3 years after study entry.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study within 4-10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed colorectal cancer meeting 1 of the following criteria:

  * Locally advanced unresectable disease
  * Distant metastatic disease
* Measurable disease
* Previously treated with at least 1, but no more than 2, prior chemotherapy regimens for unresectable locally advanced or metastatic disease

  * May have included irinotecan or oxaliplatin
  * No more than 1 prior chemotherapy regimen (not oxaliplatin-based) for advanced or metastatic disease if previously treated with oxaliplatin-based adjuvant chemotherapy
  * No more than 1 prior chemotherapy regimen (not irinotecan-based) for advanced or metastatic disease if previously treated with irinotecan-based adjuvant chemotherapy
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ upper limit of normal (ULN)
* SGOT and SGPT ≤ 2.5 times ULN

Renal

* Creatinine ≤ ULN

Cardiovascular

* No New York Heart Association class III or IV congestive heart failure
* No myocardial infarction within the past year
* No uncontrolled dysrhythmias
* No poorly controlled angina
* No prior serious ventricular arrhythmia (e.g., ventricular tachycardia or ventricular fibrillation ≥ 3 beats in a row)
* No left ventricular hypertrophy
* QTc < 500 msec
* No other significant cardiac disease

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to FR901228

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent anticancer immunotherapy

Chemotherapy

* See Disease Characteristics
* At least 28 days since prior chemotherapy and recovered
* No prior FR901228 (depsipeptide)
* No other concurrent anticancer chemotherapy

Endocrine therapy

* No concurrent anticancer hormonal therapy

Radiotherapy

* At least 28 days since prior radiotherapy and recovered
* No concurrent anticancer radiotherapy

Surgery

* At least 28 days since prior surgery and recovered

Other

* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent agent that causes QTc prolongation
* No concurrent hydrochlorothiazide
* No other concurrent investigational agents
* No other concurrent drugs that have histone deacetylase inhibitor activity (e.g., valproic acid)
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-04; Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert P. Whitehead, MD — University of Texas
Locations (88):
- United States (88):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Veterans Affairs Medical Center - Loma Linda (Pettis), Loma Linda, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago Westside Hospital, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Health System, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - University of Tennessee Cancer Institute at Methodist Central Hospital, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Veterans Affairs Medical Center - Amarillo, Amarillo, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - Sentara Cancer Institute at Sentara Norfolk General Hospital, Norfolk, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - Puget Sound Oncology Consortium, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Result] Whitehead RP, Rankin C, Hoff PM, Gold PJ, Billingsley KG, Chapman RA, Wong L, Ward JH, Abbruzzese JL, Blanke CD. Phase II trial of romidepsin (NSC-630176) in previously treated colorectal cancer patients with advanced disease: a Southwest Oncology Group study (S0336). Invest New Drugs. 2009 Oct;27(5):469-75. doi: 10.1007/s10637-008-9190-8. Epub 2008 Oct 22. PMID 18941712
- [Result] Whitehead RP, McCoy S, Wollner IS, et al.: Phase II trial of depsipeptide (NSC-630176) in colorectal cancer patients who have received either one or two prior chemotherapy regimens for metastatic or locally advanced, unresectable disease: a Southwest Oncology Group study. [Abstract] American Society of Clinical Oncology 2006 Gastrointestinal Cancers Symposium, 26-28 January 2006, San Francisco, California. A-255, 2006.